CLINICAL TRIAL: NCT06689241
Title: Rivaroxaban Versus Enoxaparin for Prophylaxis of Venous Thromboembolism in Morbidly Obese Patients Undergoing Bariatric Surgery: An open_label Randomized Controlled Trial
Brief Title: Rivaroxaban Versus Enoxaparin for Prophylaxis of Venous Thromboembolism in Bariatric Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, sarah mohamed, Lecturer anesthesia and intensive care, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0306920
Record Dates: First submitted 2024-11-13; First posted 2024-11-14 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2024-11

CONDITIONS: Morbid Obesity; Bariatric Surgery Candidate
Keywords: venous thromboembolism; enoxaparin; rivaroxaban
MeSH Terms: conditions — Obesity, Morbid; Venous Thromboembolism | interventions — Enoxaparin; Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group E (Active Comparator): 81 patients will receive subcutaneous enoxaparin 40 mg every 24 hours starting 12 hours after bariatric surgery for 14 days.
  Interventions: Drug: Enoxaparin
- group R (Experimental): 81 patients will receive oral rivaroxaban 10 mg once daily starting 24 hours after bariatric surgery for 14 days.
  Interventions: Drug: rivaroxaban

INTERVENTIONS:
Drug: Enoxaparin — 40mg
  Other Names: group E
  Arms: group E
Drug: rivaroxaban — 10mg
  Other Names: group R
  Arms: group R

SUMMARY:
Rivaroxaban versus enoxaparin for prophylaxis of venous thromboembolism in morbidly obese patients undergoing bariatric surgery: An open_label randomized controlled trial

DETAILED DESCRIPTION:
Obesity is a public health issue that raises the risk of various diseases, including diabetes, cancer, gastrointestinal disorders, depression, atherosclerotic cardiovascular disease, hypertension, and venous thromboembolism (VTE).(1) Obesity increases the risk of pulmonary embolism, a major public health concern that has been investigated since 1927.(2) Within the previous three decades, the prevalence of obesity has tripled, and surgical approaches to reduce the incidence of obesity have been studied.(3) The World Obesity Atlas 2022 predicts that by 2030, one billion people would be obese, with one in every five women and one in every seven males.(4) Over the last two decades, bariatric surgery has reduced the risk of life-threatening weight-related health issues in the United States and elsewhere.(5) Nevertheless, bariatric surgery is not without problems and is associated with a mortality rate ranging from 0.1% to 1.1.(6) Although bariatric surgery is minimally invasive, it can cause post-operative problems like dumping syndrome, anastomic leakages, malnutrition, VTE, and sepsis.(7) VTE is a leading cause of post-discharge mortality following bariatric surgery.(8) Following bariatric surgery, the incidence of postdischarge VTE was 0.29% over the course of 30 days. Despite the fact that the incidence of VTE following bariatric surgery is not particularly high, it remains the most significant cause of postdischarge mortality, in addition to the increasing incidence of obesity.(9)

Thromboprophylaxis is the primary approach to reducing VTE-induced mortality following bariatric surgery.(10) The recommended duration of VTE prevention following BS is between 7 days and 4 weeks.(11) Low-molecular-weight heparin (Enoxaparin) is used to treat and prevent deep vein thrombosis and embolism during pregnancy and after certain surgeries such as SG and RYGB. Rivaroxaban is an oral drug that directly inhibits Factor Xa, providing an alternate treatment option. Rivaroxaban is quickly absorbed and reaches peak plasma concentrations within two to four hours after intake. Rivaroxaban exhibits exceptional oral bioavailability, with absorption rates ranging from 80% to 100% for a 10 mg dose, and is not influenced by food consumption.(12)

There is paucity in the studies that evaluate the outcome of use of different thromboprophylaxis medications among patients undergoing laparoscopic sleeve gastrectomy. So this study aims to compare the effect of use of prophylactic dose of rivaroxaban 10 mg once daily and enoxaparin 40 mg every 24 hours for 14 days against the development of VTE after bariatric surgery.

Aim of the work:

The present study aims to compare the effect of use of prophylactic dose of rivaroxaban 10 mg once daily and enoxaparin 40 mg every 24 hours for 14 days against the development of VTE after bariatric surgery.

Primary outcome:

• Incidence of thromboembolic events (deep vein thrombosis, pulmonary thromboembolism, mesenteric vascular occlusion).

Secondary outcomes:

* Postoperative bleeding (hematemesis, melena).
* Length of hospital stay
* Readmission
* Reoperation

Patients :

Study settings:

This study will be conducted in general surgery department, Alexandria university hospitals.

Study design:

Open_label, randomized, prospective and controlled study Sample size calculation:(13) Based on pilot study to compare the incidence of symptomatic postoperative VTE between enoxaparin and rivaroxaban, we would need a minimum sample size of 162 patients (81 in each group) to reliably detect an effect size of δ ≥ 0.443, assuming a two-sided criterion for detection that allows for a maximum type I error rate of a= 0.05 that achieve 80% power. An expected loss to follow-up rate of 10 %, we require more patients to avoid attrition bias.

Study population:

All patients will be randomized 1:1 using a sealed envelope method. Patients will be divided into two equal groups:

Group E: 81 patients will receive subcutaneous enoxaparin 40 mg every 24 hours starting 12 hours after bariatric surgery for 14 days.

Group R: 81 patients will receive oral rivaroxaban 10 mg once daily starting 24 hours after bariatric surgery for 14 days.

Inclusion criteria:

1. Age: 20-60 years, both sexes.
2. ASA physical status class I to III.
3. BMI 35-50 kg/m²

Exclusion criteria:

1. Severe cardiac disorder
2. chronic renal failure
3. liver cirrhosis
4. major psychological disorder

Methods:

Preoperative evaluation and preparation:

* During preoperative visit, evaluation of patients will be carried out through proper history taking, clinical examination and routine laboratory investigations including complete blood picture, coagulation profile, blood urea, serum creatinine, serum electrolytes, fasting blood glucose, glycosylated hemoglobin (HBA1C), liver function tests, electrocardiogram, echocardiography and any other investigation needed.
* Patients will be informed about the need for thromboprophylaxis and the possible complications of of drugs used.
* Patients in group E will receive prophylactic dose of 40 mg of enoxaparin subcutaneously 12 hours prior to surgery, while patients in group R will receive rivaroxaban 10mg orally 24 hours before surgery.

Pre-anesthetic preparation and premedication:

* Informed written consent, from all individual participants who will be included in this study will be taken during preoperative visit.
* Elastic compression class I, knee-high type (15-18 mmHg) will be used in all patients (except in lymphedema and peripheral vascular disease).
* On arrival to operative theatre, intravenous cannula will be inserted and standard monitoring will be established using multichannel monitor (Carescape Monitor B650, GE Healthcare Finland) to monitor the following in both groups:
* Electrocardiogram (ECG) for heart rate and rhythm. (Beats/min).
* Non-invasive measurement of arterial blood pressure. (Mean blood pressure in mmHg).
* Pulse oxygen saturation. (SpO2%).
* End tidal CO2 tension (in mmHg).
* Entropy

Anesthesia:

* After preoxygenation for 3 minutes, anesthesia will be induced in both groups with propofol 2mg/kg of lean body weight until loss of verbal response, fentanyl 2µg/kg and atracurium 0.5 mg/kg intravenously. Anesthesia will be maintained by isoflurane with 50% oxygen in air (1.2-1.5 %) to maintain entropy between 40-60. Mechanical ventilation will be performed with tidal volume of 8 ml/ kg and a respiratory rate of 12-15 cycles/min to maintain the end-tidal carbon dioxide tension between 35 and 40 mmHg and an oxygen saturation of ≥ 98 per cent with 50 percent oxygen in air. Incremental doses of atracurium will be given every 30 minutes to maintain muscle relaxation.
* Intravenous dexamethasone 8 mg and ondansetron 8 mg will be given after induction for prophylaxis of postoperative nausea and vomiting.
* Multimodal analgesic techniques including 1 g of intravenous paracetamol, 0.5 mg / kg of intravenous ketorolac and pre-incisional laparoscopic preperitoneal local anesthetic infiltration to facilitate adequate pain control and early ambulation.
* Goal directed fluid therapy using pleth variability index Masimo to maintain good hydration.

At the end of surgery, awake extubation, in a semi-sitting position, will be done. Then, the patient will be transferred to the PACU.

Postoperative care:

* All patients will start clear fluids 6 hours after end of surgery.
* Early ambulation within 4-6 hours postsurgery.
* Patients in group E will receive subcutaneous enoxaparin 40 mg every 24 hours starting 12 hours after surgery for 14 days, while patients in group R will receive oral rivaroxaban 10 mg every 24 hours starting 24 hours after end of surgery for 14 days.
* All patients will be discharged home 24 hours after surgery after drain removal.
* All patients will be observed for occurrence of minor or major bleeding, deep venous thrombosis, pulmonary thromboembolism and mesenteric vascular occlusion for a period of three months after surgery.

Measurements:

The following data will be measured:

I- Demographic data:

• Patient's age (years), sex, body mass index (BMI) (kg/m2), additional VTE risk factors and co-morbidities will be recorded.

II- type and duration of surgery III- incidence of deep vein thrombosis Symptoms: calf pain Duplex ultrasonography for the legs shows DVT

IV- incidence of pulmonary thromboembolism:

Symptoms: shortness of breath, back pain, chest pain , palpitation , light headedness and syncope Signs: tachycardia, tachypnea, hypotension and cyanosis Elevated D-dimer levels, Mcconnell's sign in echocardiography and filling defects in lobar and segmental vessels in CT pulmonary angiography

V- Incidence of mesenteric vascular occlusion:

Symptoms: abdominal pain, nausea, vomiting, diarrhea and rectal bleeding. Signs: tachycardia, fever and diffuse abdominal tenderness CT angiography: thrombus in mesenteric arteries and veins, abnormal bowel wall enhancement and embolism or infarction of other organs

VI- Incidence of postoperative bleeding:

Bleeding is considered severe if it is associated with a decrease in hemoglobin of ≥ 2 g/dL compared with baseline or requiring transfusion or reoperation. All other bleeding events are considered to be minor VII- length of hospital stay (days) VIII- Incidence of reoperation IX- Incidence of readmission

X- Patient satisfaction using likert scale:

1: extremely dissatisfied, 2: dissatisfied, 3: neutral, 4: satisfied, and 5: extremely satisfied

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-60 years, both sexes.
* ASA physical status class I to III.
* BMI 35-50 kg/m²

Exclusion Criteria:

* Severe cardiac disorder
* chronic renal failure
* liver cirrhosis
* major psychological disorder

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of thromboembolic events | month 3 postoperative
  deep vein thrombosis, pulmonary thromboembolism, mesenteric vascular occlusion

SECONDARY OUTCOMES:
incidence of postoperative bleeding | one month postoperative
  hematemisis, melena
incidence of reoperation | month 3 postoperative
  number
incidence of readmission | month 3 postoperative
  number
patient satisfaction using likert scale | month 3 postoperative
  1: extremely dissatisfied, 2: dissatisfied, 3: neutral, 4: satisfied, and 5: extremely satisfied
  1: extremely dissatisfied, 2: dissatisfied, 3: neutral, 4: satisfied, and 5: extremely satisfied
  1: extremely dissatisfied, 2: dissatisfied, 3: neutral, 4: satisfied, and 5: extremely satisfied

CONTACTS AND LOCATIONS:
Overall Officials: sarah m elgamal, MD, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner J, Wruck H, Lautenbach A, von Kroge P, Wolter S, Mann O, Izbicki J, Dupree A. Comparison of Anti-factor Xa Levels in Female and Male Patients with Obesity After Enoxaparin Application for Thromboprophylaxis. Obes Surg. 2022 Mar;32(3):861-867. doi: 10.1007/s11695-021-05875-z. Epub 2022 Jan 5. PMID 34988894